CLINICAL TRIAL: NCT01289626
Title: Evaluation of Efficacy of Lanthanum Carbonate (Fosrenol) in Patients With Calciphylaxis
Brief Title: Efficacy of Lanthanum Carbonate in Calciphylaxis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2010-0127
Record Dates: First submitted 2011-02-02; First posted 2011-02-04 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Calciphylaxis
Keywords: Calciphylaxis, dialysis
MeSH Terms: conditions — Calciphylaxis | interventions — lanthanum carbonate; Lanthanum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lanthanum carbonate — FOSRENOL® will be administered orally in a dose of 1500- 3750 mg daily in divided doses with meals. Dose escalation will be utilized to a target dose of 3750 mg daily or as designated by clinician over a 4-week period from start of study. The drug will be administered for 12 weeks.
Drug: Lanthanum for calciphylaxis — Lanthanum use in calciphylaxis

SUMMARY:
The research question and primary aim is to determine if lanthanum carbonate is effective in treating calciphylaxis by measurement of complete or partial remission of skin lesions. Secondary endpoints will be measured to determine if lanthanum carbonate can lower calcium-phosphorus product levels, intact PTH and mortality. Albumin levels will be measured as a marker of nutritional status and inflammation.

DETAILED DESCRIPTION:
Calciphylaxis or calcific uremic arteriolopathy is an infrequently occurring although debilitating vasculopathy seen primarily in patients with end stage renal disease (ESRD) which almost always affects the skin. It has a prevalence rate ~4 % in long term hemodialysis patients, with 1-year survival of 45% and an 8-fold risk of death as compared to the general dialysis population. (Surgery 1997;122:1083-1089, Kidney Int 2001;60:324-332). Despite being described in the literature for over 100 years, there has been no proven effective therapy. Lanthanum carbonate (FOSRENOL®) is a potent non-aluminum, non-calcium phosphate binder that was approved for use to reduce serum phosphate levels in patients with end stage renal disease. Since the proposed etiologic mechanism of injury and vascular calcification of calciphylaxis is predominantly hyperphosphatemia, elevated serum PTH, and hypercalcemia, FOSRENOL® would be an ideal pharmacologic agent to utilize in this extremely enigmatic disease (Dermatol Clin. 2008 Oct;26(4):557-68). Furthermore, a recent case report demonstrated a significant improvement in laboratory parameters and calciphylaxis skin lesions with the use of FOSRENOL® (WMJ. 2008 Nov;107(7):335-8). The primary hypothesis is that since calciphylaxis represents the ultimate sequelae of metastatic vascular calcification predominantly involving hyperphosphatemia, elevated serum PTH, and hypercalcemia, FOSRENOL® will be efficacious in its treatment.

ELIGIBILITY:
Inclusion Criteria:

* i Participants will have signed a witnessed informed consent. ii Participants will be greater than or equal to 18 years of age iii Chronic renal failure receiving hemodialysis or peritoneal dialysis iv A diagnosis of calciphylaxis proven by skin biopsy or initial dermatology visit within the previous 5 year v Serum phosphorus > 4.5 mg/dL

Exclusion Criteria:

* i Participants are not able to understand or provide written informed consent ii The research team deems that the participant may not be able to follow the study protocol.

iii Non-dependent HD patients receiving dialysis while in acute kidney injury; iv Pregnant dialysis patient v Active gastrointestinal obstruction or bleed vi Active inflammatory bowel disease vii Acute arteriovenous graft occlusion viii Known hypersensitivity to FOSRENOL®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Remission of calciphylaxis skin lesions | 12 weeks
  The primary aim of this study will be the complete or partial remission of calciphylaxis skin lesions after 12 weeks of therapy as defined by the clinician.

SECONDARY OUTCOMES:
Measurement of phosphorus | 12 weeks
  Improvement in phosphorous control (target concentrations of 3.5 - 5.5 mg/dL) will also be monitored to correlate the relationship between phosphorous levels and calciphylaxis.
Intact PTH | 12 weeks
  Secondary aim will be the control of laboratory parameters of intact PTH
Albumin | 12 weeks
  Secondary aim will be the control of laboratory parameters of albumin
Quality of life | 12 weeks
  Demonstration of improved DLQI (Dermatology Life Quality Index, http://www.dermatology.org.uk/quality/quality-dlqi-questionnaire.html) scores

CONTACTS AND LOCATIONS:
Overall Officials: Micah Chan, MD MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospitals, Madison, Wisconsin, United States